CLINICAL TRIAL: NCT02614807
Title: Thiazide Diuretic-caused Hyponatremia in the Elderly Hypertensive: Will a Bottle of Nepro a Day Keep Hyponatremia and the Doctor Away? A Proof-of-Concept Trial
Brief Title: Protein Supplementation in Thiazide-induced Hyponatremia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult Recruitment
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201504516
Record Dates: First submitted 2015-10-21; First posted 2015-11-25 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Hyponatremia; Hypertension; Blood Pressure
Keywords: Dietary Supplement
MeSH Terms: conditions — Hyponatremia; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): All recruited patients will receive a standard endorsement of lower fluid intake (<1.5 Litres/day) by a hypertension nurse and physician and an additional treatment consisting of a bottle (237 ml) of Nepro (a low sodium, low potassium content protein supplement) a day (supply for 4 weeks will be provided).
  Interventions: Dietary Supplement: Nepro

INTERVENTIONS:
Dietary Supplement: Nepro — The intervention is a dietary protein supplement. In the elderly hypertensive patient (assuming body weight of 70 kg) with mild to moderate hyponatremia free water excess is around 2.5 L. One bottle of Nepro/day will generate about 120 mosm to be excreted via urine. Given limited and mostly fixed urinary dilution and concentration between 300 and 800 mosm/L in the elderly and very elderly, one bottle of Nepro a day will result in an extra 400 ml of urine for a net loss of 163 ml of free water. Thus over the period of 2 to 4 weeks the calculated free water excess should be completely eliminated.

SUMMARY:
High blood pressure is very common among elderly Canadians. Clinical trials show clear benefit from lowering blood pressure in hypertensive elderly patients. These trials also demonstrate safety for several classes of blood pressure lowering drugs including water pills. However, water pills (thiazide diuretics) used for treatment of hypertension, can cause low sodium (hyponatremia), a significant clinical problem mainly among elderly and very elderly. Causes are age related decrease in kidneys' ability to get rid of water and low salt coupled with high water intake. A standard approach to treatment is lacking since higher salt intake may worsen hypertension, and lower water and higher protein intake is difficult to understand and actually implement. 'Nepro' is a nutritional drink high in protein, and low in potassium and sodium. It is used frequently as a dietary supplement in patients with kidney disease specifically for low sodium and high protein content. The high protein content in Nepro can help the kidney get rid of excess water, and the low sodium and potassium content will make this a safe option to use. Hence investigators propose a proof-of-concept trial on an easy to understand and administer, and relatively affordable solution to this issue. It could be summarized in one sentence: "Will a bottle of Nepro a day keep thiazide-caused hyponatremia and the doctor away?"

ELIGIBILITY:
Inclusion Criteria:

* Elderly (>65 years old)
* with diagnosed hypertension (HTN) treated with thiazide (hydrochlorothiazide) or thiazide-like (chlorthalidone and indapamide) diuretic and
* mild to moderate hyponatremia (Plasma sodium concentration 125-133 mmol/L).

Exclusion Criteria:

* Pregnancy
* estimated glomerular filtration rate (eGFR) <45 ml/min/1.75 m2,
* Other causes of hyponatremia (liver cirrhosis, uncontrolled hypothyroidism, adrenal insufficiency)
* unable to provide informed consent;
* patients with generalized volume overload who may require immediate changes in diuretic therapy (at the discretion of treating HTN specialist);
* patients taking drugs which may interfere with urinary sodium excretion (such as carbamazepine, loop diuretics, potassium sparing diuretics, mineralocorticoid and glucocorticosteroids, selective serotonin receptor inhibitors, tricyclic antidepressants, amiodarone, and lithium);
* patients with moderate to severe hyponatremia (Plasma sodium concentration < 125 mmol/L) who may require immediate discontinuation of the thiazide diuretic .

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: Correction of Hyponatremia (Serum Sodium > 133 mmol/L or reduction of deficit by 50%) | 4 weeks
  The cumulative proportion of participants whose serum sodium either normalizes (>133 mmol/L) by 4 weeks or who exhibit a decrease in deficit by 50% compared to baseline level.

SECONDARY OUTCOMES:
Feasibility: recruitment (proportion of patients who are screened and eligible, and proportion eligible who consent) | 4 weeks
  The proportion of patients who are screened and found to be eligible and the proportion of those eligible who actually consent for the study
Safety: Tolerability of intervention (proportion of patients who can tolerate the Nepro supplement) | 2 and 4 weeks
  The proportion of patients who tolerate the Nepro supplement for the duration of the study, and who are able to comply with the daily supplementation for the period of study.
Safety: Worsening of hyponatremia (proportion of patients with Sodium < 125 mmol/L at 2 or 4 weeks) | 2 and 4 weeks
  In addition, the proportion of patients who might have a worsening of hyponatremia (plasma sodium < 125 mmol/L) either at 2 weeks or at 4 weeks, which will result in immediate discontinuation of the thiazide diuretic will also be measured and reported

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Ruzicka, MD PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruzicka M, McCormick B, Magner P, Ramsay T, Edwards C, Bugeja A, Hiremath S. Thiazide diuretic-caused hyponatremia in the elderly hypertensive: will a bottle of Nepro a day keep hyponatremia and the doctor away? Study protocol for a proof-of-concept feasibility trial. Pilot Feasibility Stud. 2018 Apr 6;4:71. doi: 10.1186/s40814-018-0263-y. eCollection 2018. PMID 29636984